CLINICAL TRIAL: NCT05179902
Title: Predictive Properties of Myocardial Fibrosis Biomarkers on the Outcome of Atrial Fibrillation Ablation
Acronym: PROFIB-AF
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University Hospital, Clermont-Ferrand (Other)
Collaborators: Groupama foundation (Unknown); Biochemistry Lab University Hospital Clermont-Ferrand (Unknown)
Responsible Party: Sponsor
Other Study IDs: RNI 2021 MASSOULIE; 2021-A02091-40 (Other: 2021-A02091-40)
Record Dates: First submitted 2021-12-17; First posted 2022-01-06 (Actual); Last update posted 2022-02-02 (Actual); Status verified 2022-02

CONDITIONS: Women and Men Over 18 Years Old; AF Ablation (ECS recommendation2020&ACS2014) Either for Paroxysmal AF Unresponsive to Anti-arrhythmic Treatment Either for Persisting Symptomatic AF; Able to Give His Non Opposition to Participate to the Study
Keywords: Atrial fibrillation (AF); Myocardial fibrosis; AF ablation; AF recurrence; Biological collection; AF and myocardial fibrosis biological markers
MeSH Terms: conditions — Atrial Fibrillation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Atrial fibrillation (AF) is the most common cardiac arrhythmia. As an independent predictor of cardiovascular mortality, particularly for stroke, its management is a real public health issue. AF is associated with diabetes, obesity, hypertension, heart failure and, occasionally, hyperthyroidism. Atrial fibrosis is one of the major players in the genesis and maintenance of AF. It has a strong impact on rhythmic prognosis and treatment success.

Currently the AF ablation is the treatment recommended by the European Society of Cardiology (ESC) and by the American Society of Cardiology. The rate of AF recurrence is variable according to the patient characteristics and remains unfortunately today difficult to predict.

Abnormal concentrations of circulating biomarkers reflecting the underlying pathophysiologic mechanisms of myocardial fibrosis could help to identify patients at higher risk of developing AF and/or AF recurrence after ablation. Thus, the development of simple, reliable and valid biological tests of atrial fibrosis would allow the clinicians i) to estimate the potential success of AF ablation; ii) to predict AF recurrence; iv) and to propose a AF personalized therapeutic approach.

The main objective of PROFIB-AF study is to identify, among biological markers (ICTP, PICP, PIIINP, sRAGE, AGE, Galectin 3, sSt2, microRNAs) of myocardial fibrosis, those which can predict the recurrence risk after AF ablation.

DETAILED DESCRIPTION:
Patients prone to AF ablation and do not object to participate at PROFIB-AF study will be offered, in parallel of their conventional care, blood samples the day of AF ablation by femoral and sinusal punctures and 12 months after ablation by venipuncture for the biomarkers analysis.

As part of their traditional care, these patients will benefit several exams beforeAF ablation (MRI, clinical examination ECG, echocardiography, routine biological analyzes), and four follow-up visits after AF ablation (at 3, 6, 9 and 12 months post-ablation) to evaluate AF recurrence, occurrence of MACE and heart failure signs.

ELIGIBILITY:
Inclusion Criteria:

* Adult patient, male or female, eligible for an AF ablation procedure according to the recommendations (European Society of Cardiology 2020 and American Society of Cardiology 2014), either for symptomatic paroxysmal AF refractory to anti-arrhythmic treatments (or in first intention according to patient preference), or for symptomatic persistent AF.
* Able to give their non-opposition to participate in the research.
* Affiliation to a social security regime.

Exclusion Criteria:

* Any pro-fibrotic phenomenon that may interfere with the interpretation of the results, i.e. severe valvular heart disease, amyloid heart disease, dilated cardiomyopathy of non-rhythmic origin, hypertrophic cardiomyopathy, severe ischaemic heart disease (late revascularisation, LV dysfunction, disturbed kinetics), COPD > stage 2, pulmonary fibrosis, renal failure > stage 3A, hepatic cirrhosis, hepatocellular failure, recent invasive surgery < 3 months
* Life expectancy less than 1 year
* Pregnant or breastfeeding women
* Patients of legal age under protective supervision (guardianship, trusteeship)
* Refusal to participate

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Major patient eligible for an AF ablation procedure according to the recommendations (European Society of Cardiology 2020 and American Society of Cardiology 2014), either for symptomatic paroxysmal AF refractory to anti-arrhythmic treatments (or in first intention according to patient preference), or for symptomatic persistent AF.
Sampling Method: Probability Sample
Enrollment: 190 (Estimated)
Dates: Start 2022-01-20 (Actual); Primary Completion 2025-01 (Estimated); Study Completion 2025-01 (Estimated)

PRIMARY OUTCOMES:
Occurrence of an atrial fibrillation recurrence | Any AF episode >30 seconds at pre-ablation (yes or no)
  ECG 12 lead profile
Occurrence of an atrial fibrillation recurrence | Any AF episode >30 seconds at 3 months (yes or no)
  ECG 12 lead profile
Occurrence of an atrial fibrillation recurrence | Any AF episode >30 seconds at 6 months (yes or no)
  ECG 12 lead profile
Occurrence of an atrial fibrillation recurrence | Any AF episode >30 seconds at 12 months (yes or no)
  ECG 12 lead profile
Occurrence of an atrial fibrillation recurrence | Any AF episode >30 seconds at pre-ablation (yes or no)
  Holter ECG
Occurrence of an atrial fibrillation recurrence | Any AF episode >30 seconds at 3 months (yes or no)
  Holter ECG
Occurrence of an atrial fibrillation recurrence | Any AF episode >30 seconds at 6 months (yes or no)
  Holter ECG
Occurrence of an atrial fibrillation recurrence | Any AF episode >30 seconds at 12 months (yes or no)
  Holter ECG
Occurrence of an atrial fibrillation recurrence | PIIINP at pre-ablation (in ng/mL
  Biological markers profil
Occurrence of an atrial fibrillation recurrence | PIIINP at 12 months (in ng/mL)
  Biological markers profil
Occurrence of an atrial fibrillation recurrence | ICTP at pre-ablation (in ng/mL)
  Biological markers profil
Occurrence of an atrial fibrillation recurrence | ICTP at 12 months (in ng/mL)
  Biological markers profil
Occurrence of an atrial fibrillation recurrence | PICP at pre-ablation (in ng/mL)
  Biological markers profil
Occurrence of an atrial fibrillation recurrence | PICP at 12 months (in ng/mL)
  Biological markers profil
Occurrence of an atrial fibrillation recurrence | sRAGE at pre-ablation (in pg/mL)
  Biological markers profil
Occurrence of an atrial fibrillation recurrence | sRAGE at 12 months (in pg/mL)
  Biological markers profil
Occurrence of an atrial fibrillation recurrence | AGE at pre-ablation (in ng/mL)
  Biological markers profil
Occurrence of an atrial fibrillation recurrence | AGE at 12 months (in ng/mL)
  Biological markers profil

SECONDARY OUTCOMES:
Rate of fibrosis of the left atrium | Degree of left atrial fibrosis on MRI at the inclusion (pre-ablation; in %)
  IRM profile
Rate of fibrosis of the left atrium | Endocardial left atria low voltage area (<0.5mV) in sinus rhythm (in %)
  Voltage mapping
Dominant frequency of AF | F wave frequency at the inclusion (pre-ablation; in ms)
  ECG 12 lead profil
Dominant frequency of AF | F wave frequency at 3 months (in ms)
  ECG 12 lead profil
Dominant frequency of AF | F wave frequency at 6 months (in ms)
  ECG 12 lead profil
Dominant frequency of AF | F wave frequency at 12 months (in ms)
  ECG 12 lead profil
Dominant frequency of AF | F wave amplitude at the inclusion (pre-ablation; in mv)
  ECG 12 lead profil
Dominant frequency of AF | F wave amplitude at 3 months (in mv)
  ECG 12 lead profil
Dominant frequency of AF | F wave amplitude at 6 months (in mv)
  ECG 12 lead profil
Dominant frequency of AF | F wave amplitude at 12 months (in mv)
  ECG 12 lead profil
Dominant frequency of AF | AF characteristics at the inclusion (pre-ablation; paroxysmal, persistent)
  ECG 12 lead profil
Dominant frequency of AF | AF characteristics at 3 months (paroxysmal, persistent)
  ECG 12 lead profil
Dominant frequency of AF | AF characteristics at 6 months (paroxysmal, persistent)
  ECG 12 lead profil
Dominant frequency of AF | AF characteristics at 12 months (paroxysmal, persistent)
  ECG 12 lead profil
Dominant frequency of AF | AF duration at the inclusion (pre-ablation, in ms)
  ECG 12 lead profil
Dominant frequency of AF | AF duration at 3 months (in ms)
  ECG 12 lead profil
Dominant frequency of AF | AF duration at 6 months (in ms)
  ECG 12 lead profil
Dominant frequency of AF | AF duration at 12 months (in ms)
  ECG 12 lead profil
Dominant frequency of AF | F wave frequency at the inclusion (pre-ablation; in ms)
  Holter ECG profil
Dominant frequency of AF | F wave frequency at 3 months (in ms)
  Holter ECG profil
Dominant frequency of AF | F wave frequency at 6 months (in ms)
  Holter ECG profil
Dominant frequency of AF | F wave frequency at 9 months (in ms)
  Holter ECG profil
Dominant frequency of AF | F wave frequency at 12 months (in ms)
  Holter ECG profil
Dominant frequency of AF | F wave amplitude at the inclusion (pre-ablation; in mV)
  Holter ECG profil
Dominant frequency of AF | F wave amplitude at 3 months (in mV)
  Holter ECG profil
Dominant frequency of AF | F wave frequency at 6 months (in mV)
  Holter ECG profil
Dominant frequency of AF | F wave amplitude at 9 months (in mV)
  Holter ECG profil
Dominant frequency of AF | F wave amplitude at 12 months (in mV)
  Holter ECG profil
Dominant frequency of AF | AF characteristics at the inclusion (pre-ablation; paroxysmal, persistent)
  Holter ECG profil
Dominant frequency of AF | AF characteristics at 3 months (paroxysmal, persistent)
  Holter ECG profil
Dominant frequency of AF | AF characteristics at 6 months (paroxysmal, persistent)
  Holter ECG profil
Dominant frequency of AF | AF characteristics at 9 months (paroxysmal, persistent)
  Holter ECG profil
Dominant frequency of AF | AF characteristics at 12 months (paroxysmal, persistent)
  Holter ECG profil
Dominant frequency of AF | AF duration at the inclusion (pre-ablation; in ms)
  Holter ECG profil
Dominant frequency of AF | AF duration at 3 months (in ms)
  Holter ECG profil
Dominant frequency of AF | AF duration at 6 months (in ms)
  Holter ECG profil
Dominant frequency of AF | AF duration at 9 months (in ms)
  Holter ECG profil
Dominant frequency of AF | AF duration at 12 months (in ms)
  Holter ECG profil
Dominant frequency of AF | Left atria volume at pre-ablation (mL)
  Echocardiography
Dominant frequency of AF | Left atria volume at 12 months (mL)
  Echocardiography
Dominant frequency of AF | Indexed left atria volume at pre-ablation (mL)
  Echocardiography
Dominant frequency of AF | Indexed left atria volume at 12 months (mL)
  Echocardiography
Dominant frequency of AF | LVEF at the inclusion (pre-ablation; %)
  Echocardiography
Dominant frequency of AF | LVEF at 12 months (%)
  Echocardiography
Dominant frequency of AF | Hemoglobin at pre-ablation (in g/dL)
  Biological profil
Dominant frequency of AF | Hemoglobin at 12 months (in g/dL)
  Biological profil
Dominant frequency of AF | HbA1c at pre-ablation (in %)
  Biological profil
Dominant frequency of AF | HbA1c at 12 months (in %)
  Biological profil
Dominant frequency of AF | Kalemia at pre-ablation (in mmol/L)
  Biological profil
Dominant frequency of AF | Kalemia at 12 months (in mmol/L)
  Biological profil
Dominant frequency of AF | Natremia at pre-ablation (in mmol/L)
  Biological profil
Dominant frequency of AF | Natremia at 12 months (in mmol/L)
  Biological profil
Dominant frequency of AF | Glycemia at pre-ablation (in mmol/L)
  Biological profil
Dominant frequency of AF | Glycemia at 12 months (in mmol/L)
  Biological profil
Dominant frequency of AF | Total bilirubin at pre-ablation (in µmol/L)
  Biological profil
Dominant frequency of AF | Total bilirubin at 12 months (in µmol/L)
  Biological profil
Dominant frequency of AF | ASAT at pre-ablation (in U/L)
  Biological profil
Dominant frequency of AF | ASAT at 12 months (in U/L)
  Biological profil
Dominant frequency of AF | ALAT at pre-ablation (in U/L)
  Biological profil
Dominant frequency of AF | ALAT at 12 months (in U/L)
  Biological profil
Dominant frequency of AF | GGT at pre-ablation (in U/L)
  Biological profil
Dominant frequency of AF | GGT at 12 months (in U/L)
  Biological profil
Dominant frequency of AF | PAL at pre-ablation (in U/L)
  Biological profil
Dominant frequency of AF | PAL at 12 months (in U/L)
  Biological profil
Dominant frequency of AF | LDH at pre-ablation (in U/L)
  Biological profil
Dominant frequency of AF | LDH at 12 months (in U/L)
  Biological profil
Dominant frequency of AF | Creatinine level at pre-ablation (in µmol/L)
  Biological profil
Dominant frequency of AF | Creatinine level at 12 months (in µmol/L)
  Biological profil
Dominant frequency of AF | Clearance CKD-EPI at pre-ablation (ml/min/1.73m²)
  Biological profil
Dominant frequency of AF | Clearance CKD-EPI at 12 months (ml/min/1.73m²)
  Biological profil
Dominant frequency of AF | Urea at pre-ablation (mmol/L)
  Biological profil
Dominant frequency of AF | Urea at 12 months (mmol/L)
  Biological profil
Dominant frequency of AF | Protidemia at pre-ablation (g/L)
  Biological profil
Dominant frequency of AF | Protidemia at 12 months (g/L)
  Biological profil
Dominant frequency of AF | NTproBNP at pre-ablation (ng/L)
  Biological profil
Dominant frequency of AF | NTproBNP at 12 months (ng/L)
  Biological profil
Dominant frequency of AF | TSH at pre-ablation (mUI/L)
  Biological profil
Dominant frequency of AF | TSH at 12 months (mUI/L)
  Biological profil
Dominant frequency of AF | T3 at pre-ablation (pmol/L)
  Biological profil
Dominant frequency of AF | T3 at 12 months (pmol/L)
  Biological profil
Dominant frequency of AF | T4 at pre-ablation (pmol/L)
  Biological profil
Dominant frequency of AF | T4 at 12 months (pmol/L)
  Biological profil
Dominant frequency of AF | Galectin-3 at pre-ablation (in ng/mL)
  Biological profil
Dominant frequency of AF | Galectin-3 at 12 months (in ng/mL)
  Biological profil
Dominant frequency of AF | sST2 at pre-ablation (in ng/mL)
  Biological profil
Dominant frequency of AF | sST2 at 12 months (in ng/mL)
  Biological profil
Dominant frequency of AF | miRNAs at pre-ablation (fold change)
  Biological profil
Dominant frequency of AF | miRNAs at 12 months (fold change)
  Biological profil
Dominant frequency of AF | Diabete at pre-ablation (yes, type I, type II or no)
  Diabete profil
Dominant frequency of AF | Body weight at pre-ablation (in kg)
  Clinical exam
Dominant frequency of AF | Body weight at 3 months (in kg)
  Clinical exam
Dominant frequency of AF | Body weight at 6 months (in kg)
  Clinical exam
Dominant frequency of AF | Body weight at 12 months (in kg)
  Clinical exam
Dominant frequency of AF | Body height at pre-ablation (in cm)
  Clinical exam
Dominant frequency of AF | Body height at 3 months (in cm)
  Clinical exam
Dominant frequency of AF | Body height at 6 months (in cm)
  Clinical exam
Dominant frequency of AF | Body height at 12 months (in cm)
  Clinical exam
Dominant frequency of AF | Systolic blood pressure at pre-ablation (in mmHg)
  Clinical exam
Dominant frequency of AF | Systolic blood pressure at 3 months (in mmHg)
  Clinical exam
Dominant frequency of AF | Systolic blood pressure at 6 months (in mmHg)
  Clinical exam
Dominant frequency of AF | Systolic blood pressure at 12 months (in mmHg)
  Clinical exam
Dominant frequency of AF | Diastolic blood pressure at pre-ablation (in mmHg)
  Clinical exam
Dominant frequency of AF | Diastolic blood pressure at 3 months (in mmHg)
  Clinical exam
Dominant frequency of AF | Diastolic blood pressure at 6 months (in mmHg)
  Clinical exam
Dominant frequency of AF | Diastolic blood pressure at 12 months (in mmHg)
  Clinical exam
Dominant frequency of AF | Cardiac frequency pressure at pre-ablation (in bpm)
  Clinical exam
Dominant frequency of AF | Cardiac frequency pressure at 3 months (in bpm)
  Clinical exam
Dominant frequency of AF | Cardiac frequency pressure at 6 months (in bpm)
  Clinical exam
Dominant frequency of AF | Cardiac frequency pressure at 12 months (in bpm)
  Clinical exam
Dominant frequency of AF | NYHA score at pre-ablation (I, II, III or IV)
  Clinical exam
Dominant frequency of AF | NYHA score at 3 months (I, II, III or IV)
  Clinical exam
Dominant frequency of AF | NYHA score at 6 months (I, II, III or IV)
  Clinical exam
Dominant frequency of AF | NYHA score at 12 months (I, II, III or IV)
  Clinical exam
Dominant frequency of AF | Congestive signs at pre-ablation (yes, left, right, global; or not)
  Clinical exam
Dominant frequency of AF | Congestive signs at at 3 months (yes, left, right, global; or not)
  Clinical exam
Dominant frequency of AF | Congestive signs at 6 months (yes, left, right, global; or not)
  Clinical exam
Dominant frequency of AF | Congestive signs at 12 months (yes, left, right, global; or not)
  Clinical exam

CONTACTS AND LOCATIONS:
Overall Officials: Grégoire Massoulié, Principal Investigator — University Hospital, Clermont-Ferrand
Locations (1):
- CHU clermont-ferrand, Clermont-Ferrand, France